CLINICAL TRIAL: NCT03578601
Title: Predictive Parameters for Difficult Tracheal Intubation Identification in Thyroid Surgery, a Observational Monocentric Prospective Study
Brief Title: Predictive Parameters for Difficult Tracheal Intubation Identification in Thyroid Surgery
Status: Completed | Type: Observational
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Alessandro De Cassai, Medical Doctor, University of Padova
Other Study IDs: 4133/AO/17
Record Dates: First submitted 2018-02-19; First posted 2018-07-06 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Intubation;Difficult
Keywords: Intubation; Difficult; thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroid surgery: Patient undergoing thyroid surgery
  Interventions: Other: Thyroid surgery

INTERVENTIONS:
Other: Thyroid surgery — Patient undergoing thyroid surgery

SUMMARY:
Intubation manoeuvres in patients undergoing thyroid surgery might be challenging for anesthesiologist. Thyroid gland enlargement (goiter) or tissue fibrosis (neoplasms) could alter the physiologic anatomy of upper airways and trachea, resulting in compression or dislocation. We want to evaluate the incidence and identify predictive parameters of difficult intubation in patients undergoing thyroid surgery.

DETAILED DESCRIPTION:
Intubation manoeuvres in patients undergoing thyroid surgery might be challenging for anesthesiologist. Thyroid gland enlargement (goiter) or tissue fibrosis (neoplasms) could alter the physiologic anatomy of upper airways and trachea, resulting in compression or dislocation.

There are few scientific data about airway management and thyroid pathology and the incidence of difficult tracheal intubation in this specific kind of patient is largely variable from 0% to 12.9%. These data have been collected from little statistical samples (from 50 to 326 patients), the results aren't always unanimous and a study evaluating simultaneously all the risk factors for difficult intubation does not exist.

We want to evaluate the incidence and identify predictive parameters of difficult intubation in patients undergoing thyroid surgery.

During pre-anesthetic assessment the following data will be collected:

Inter-incisor gap (cm) Mallampati test (1;2;3;4) Thyromental distance (cm) Prognathism (yes; no) Neck motility (<80°;80-90°;>90°) Total body weight (kg) History of difficult tracheal intubation (yes; no) Tracheal deviation at chest X-Ray (yes; no) Neck circumference (cm) Mediastinal goiter (yes; no) Histologic features (benign; carcinoma)

During the post-anesthesia it will be noted down the following:

Cormack scale (1; 2a; 2b; 3; 4) Number of necessary attempts to intubate (1;2;3;…) Time from induction to intubation (min) Necessity to use advanced airway management devices (Frova; Glidescope; Ambu-scope; fiber-optic; other)

ELIGIBILITY:
Inclusion Criteria:

* thyroid surgery

Exclusion Criteria:

* <18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-17 (Actual); Study Completion 2018-09-17 (Actual)

PRIMARY OUTCOMES:
Difficult intubation incidence | through study completion, an average of 2 year
  Difficult intubation described as Cormack 3 or 4

SECONDARY OUTCOMES:
Histologic features (benign; carcinoma) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Histologic features (benign; carcinoma) as predictive parameter for difficult intubation
Neck circumference (cm) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Neck circumference (cm) as predictive parameter for difficult intubation
Tracheal deviation at chest X-Ray (yes; no) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Tracheal deviation at chest X-Ray (yes; no) as predictive parameter for difficult intubation
History of difficult tracheal intubation (yes; no) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative History of difficult tracheal intubation (yes; no) as predictive parameter for difficult intubation
Total body weight (kg) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Total body weight (kg) as predictive parameter for difficult intubation
Neck motility (<80°;80-90°;>90°) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Neck motility (<80°;80-90°;>90°) as predictive parameter for difficult intubation
Thyromental distance (cm) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Thyromental distance (cm) as predictive parameter for difficult intubation
Mediastinal goiter (yes; no) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Mediastinal goiter (yes; no) as predictive parameter for difficult intubation
Prognathism (yes; no) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Prognathism (yes; no) as predictive parameter for difficult intubation
Mallampati test (1;2;3;4) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Mallampati test (1;2;3;4) as predictive parameter for difficult intubation
Inter-incisor gap (cm) as predictive parameter for difficult intubation | through study completion, an average of 2 year
  preoperative Inter-incisor gap (cm) as predictive parameter for difficult intubation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Probably all IPD will be shared at the end of the study

REFERENCES:
- [Background] Petrini F, Accorsi A, Adrario E, Agro F, Amicucci G, Antonelli M, Azzeri F, Baroncini S, Bettelli G, Cafaggi C, Cattano D, Chinelli E, Corbanese U, Corso R, Della Puppa A, Di Filippo A, Facco E, Favaro R, Favero R, Frova G, Giunta F, Giurati G, Giusti F, Guarino A, Iannuzzi E, Ivani G, Mazzon D, Menarini M, Merli G, Mondello E, Muttini S, Nardi G, Pigna A, Pittoni G, Ripamonti D, Rosa G, Rosi R, Salvo I, Sarti A, Serafini G, Servadio G, Sgandurra A, Sorbello M, Tana F, Tufano R, Vesconi S, Villani A, Zauli M; Gruppo di Studio SIAARTI "Vie Aeree Difficili"; IRC e SARNePI; Task Force. Recommendations for airway control and difficult airway management. Minerva Anestesiol. 2005 Nov;71(11):617-57. No abstract available. English, Italian. PMID 16278626
- [Background] Frova G, Sorbello M. Algorithms for difficult airway management: a review. Minerva Anestesiol. 2009 Apr;75(4):201-9. Epub 2008 Oct 23. PMID 18946426
- [Result] Bouaggad A, Nejmi SE, Bouderka MA, Abbassi O. Prediction of difficult tracheal intubation in thyroid surgery. Anesth Analg. 2004 Aug;99(2):603-6, table of contents. doi: 10.1213/01.ANE.0000122634.69923.67. PMID 15271749
- [Result] Amathieu R, Smail N, Catineau J, Poloujadoff MP, Samii K, Adnet F. Difficult intubation in thyroid surgery: myth or reality? Anesth Analg. 2006 Oct;103(4):965-8. doi: 10.1213/01.ane.0000237305.02465.ee. PMID 17000813
- [Result] Meco BC, Alanoglu Z, Yilmaz AA, Basaran C, Alkis N, Demirer S, Cuhruk H. Does ultrasonographic volume of the thyroid gland correlate with difficult intubation? An observational study. Braz J Anesthesiol. 2015 May-Jun;65(3):230-4. doi: 10.1016/j.bjane.2014.06.004. Epub 2014 Oct 16. PMID 25925037
- [Result] Khan MN, Rabbani MZ, Qureshi R, Zubair M, Zafar MJ. The predictors of difficult tracheal intubations in patients undergoing thyroid surgery for euthyroid goitre. J Pak Med Assoc. 2010 Sep;60(9):736-8. PMID 21381580